CLINICAL TRIAL: NCT06650436
Title: DEliriuM in STroke: the Link Between Stroke, Delirium and Long-term Cognitive Impairment
Acronym: DE-MIST
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel (Other); UMC Utrecht (Other)
Responsible Party: Principal Investigator, Fenne Vandervorst, Principal Investigator, Universitair Ziekenhuis Brussel
Other Study IDs: 23375_DE_MIST
Record Dates: First submitted 2024-05-13; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Ischemic Stroke; Delirium; Cognitive Impairment
Keywords: Post stroke delirium; Post-stroke cognitive impairment; EEG; Delirium; Ischemic Stroke; Cognitive Impairment
MeSH Terms: conditions — Ischemic Stroke; Delirium; Cognitive Dysfunction | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- no delirium post-stroke
  Interventions: Diagnostic Test: EEG; Diagnostic Test: MRI; Diagnostic Test: Depression screening and neuropsychological tests
- post-stroke delirium
  Interventions: Diagnostic Test: EEG; Diagnostic Test: MRI; Diagnostic Test: Depression screening and neuropsychological tests

INTERVENTIONS:
Diagnostic Test: EEG — The phase lag index will be used to assess functional connectivity between time series based on the consistency with which one signal is leading or lagging with respect to another signal.The PLI characterizes the asymmetry in the distribution of instantaneous phase differences between signals. If such an asymmetry is present, a phase coupling is assumed between signals, reflecting synchronized activity. Importantly, zero-phase coupling is discarded in the PLI as this may represent activity from common sources picked up at different electrodes. Based on the MST, network measures can be calculated. It is a measure of network efficiency. Leaf fraction quantifies the fraction of nodes in the whole network that have only one connecting edge, which is a measure of network integration.
Diagnostic Test: MRI — Manual segmentation of the acute ischemic lesion will be performed on MRI of the brain. Support vector regression-based lesion symptom mapping (SVR-LSM) will be performed to determine the association between AIL location and PSD. We will also perform an assumption-free region of interest (ROI)-based analysis by using support vector regression. The ROIs will be determined by the AAL atlas and ICBM-DTI-81 white matter tract atlas in MNI-152 space.
  The MRI's will be performed within 72 hours of the stroke onset with a follow-up of 12 months.
Diagnostic Test: Depression screening and neuropsychological tests — Screening post-stroke delirium (during first 72hours after stroke symptom onset):
  4AT test score: 0-12 (>/= 4: diagnosis of (post-stroke) delirium) RASS score: from -5 until +4 Screening post-stroke cognitive impairment (3months, 12 months): MOCA score: 0-30
  Screening post-stroke depression:
  Patient Health Questionnaire-2: score 0-6 Hospital Anxiety and Depression Scale: score 0-21Anxiety and 0-21Depression

SUMMARY:
Primary objective of this study:

determine whether PSD is a risk factor for PSCI, independent of brain frailty and premorbid cognitive functioning.

Secondary objectives:

1. to investigate the role of infarct location, imaging markers of brain frailty and brain network disintegration in the development of PSD;
2. to investigate the role of persistent brain network disintegration in the development of PSCI.

DETAILED DESCRIPTION:
1. Patient characteristics such as age, (premorbid) modified Rankin Scale (mRS) and stroke characteristics such as stroke severity (NIHSS) will be documented. There will be screened for preexisting cognitive decline (by using a Dutch shortened and validated version of the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE). Clinical assessments such as NIHSS and mRS will be repeated after 3 and 12 months, as part of regular care. Comorbid conditions will be documented during the whole duration of the study.
2. Previous or concomitant use of drugs will be registered, in particular those known to affect cognitive function, such as anticholinergic drugs, analgo-sedatives or benzodiazepines.
3. Delirium assessment during hospitalization: delirium assessment will be performed twice a day, at the beginning and ending of each day shift with a minimal interval of 5 hours between the two evaluations each day, during the first 72 hours after ischemic stroke onset. The length of the screening period is based on the results of a prospective observational study that showed that almost all of PSD cases occurred within 72 hours (98%). If a patient develops delirium during the first 72 hours after stroke onset, delirium monitoring will be continued until 4 negative screening tests are obtained (because of possible fluctuations of delirium signs) or until the end of the hospitalization. Delirium assessments will be performed by a trained nurse using the 4 'A's Test (4AT) and the Richmond Agitation and Sedation Scale (RASS). The RASS will be used to determine the type of delirium, with negative RASS scores indicating hypoactive delirium and a positive RASS score indicating hyperactive delirium.
4. EEG recordings will be performed by a trained neurophysiology nurse, using 21 electrodes placed according to the 10-20 system, with 10 minutes eyes open and 10 minutes eyes closed, within one hour of the clinical evaluation during the hospitalization. The first EEG will be routinely recorded during the first 24 hours after stroke onset. A second EEG will be only be recorded in patients who develop PSD between 24 and 72 hours after stroke onset. EEG's recorded during hospitalization are considered standard of care. EEG recording will be repeated at 12 months.
5. MRI of the brain will be performed during hospitalization (=standard of care) and 12 months after stroke onset. Standard acute stroke imaging will involve a 3-T MR scanner with sagittal 3DFLAIR (fluid-attenuated inversion recovery) sequence, T2 sequence fossa posterior with a slice thickness of 2mm, axial diffusion sequence (slice thickness 4mm), 3D-SWI (susceptibility weighted imaging) sequence (slice thickness 2mm) and 3D-QALAS sequence. Manual segmentation of the acute ischemic lesion will be performed on MRI scans of the brain, performed during hospitalization for IS. Patients without visible acute ischemic lesions on MRI will be excluded. Acute ischemic stroke lesions (AIL) are defined by the presence of a hyperintense MRI diffusion-weighted imaging (DWI) lesion with corresponding hypointensity in apparent diffusion coefficient map (ADC). The DWI and ADC images may also help to discriminate between new ischemic lesions and pre-existent white matter hyperintensities. Prior to performing the segmentations for the current study, the reviewer will delineate AIL on 10 scans twice with an interval of 1 month, with the aim to optimize intraobserver agreement. Visual rating of white matter hyperintensities (Fazekas scale) and cerebral atrophy (global cortical atrophy (GCA) scale) as markers of brain frailty.
6. Cognitive and mood assessment: neuropsychological assessment will take place at 3 months and 12 months after the IS. A trained nurse will administer the Montreal Cognitive Assessment (MOCA, Dutch or French version) at these time intervals. She will be blinded for the initial occurrence of delirium. Depression screening will be performed at the same time intervals by using the Patient Health Questionnaire-2 and the Hospital Anxiety and Depression Scale (HADS) (in order to be able to compare with previously performed delirium studies).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* clinical diagnosis of first-ever ischemic stroke (onset <72h at time of inclusion),
* admitted at stroke unit of UZ Brussel,
* ability to participate in cognitive assessments,
* fluency in Dutch or French,
* ability to undergo an EEG during the first 24 hours after onset of stroke symptoms,
* ability to undergo MRI of the brain.

Exclusion Criteria:

* epilepsy history,
* pre-existing, space occupying brain lesion (except small meningeoma),
* pregnancy or wish to become pregnant,
* severe language impairment or dementia impeding cognitive assessment, life expectancy of less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized at the stroke unit of UZ Brussel, who can be included within 72 hours after stroke symptom onset.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Post-stroke delirium | first 72 hours after stroke symptom onset
  Firstly using the 4 A's test (4AT) to screen for delirium. This score can go from 0 which indicates no suspicion of delirium; to a score higher than 4 which does indicates a higher suspicion of delirium. Then we'll further analyse the type of delirium using the Richmond Agitation-Sedation Scale (RASS). This scale has 2 types of scores, the first one being the negative scores (-5 -> -1) that fits a hypoactive presentation of delirium. 0 is a normal score, indicating an alert and calm patient. The positive scores (1 -> 4) are administered in case of hyperactive presentations of delirium.
The role of brain network disintegration in post-stroke delirium: electrical analysis of the relative power in the alfa frequency band | first 72 hours after stroke symptom onset
  To further understand the underlying brain activity during post-stroke delirium we'll perform an additional electroencephalogram (EEG) to look at potential deviations in the brain activity that could be connected to this clinical presentation. We'll specifically look at the relative power in the alfa frequency band.
The role of brain network disintegration in post-stroke delirium: electrical analysis of the relative power in the beta frequency band | first 72 hours after stroke symptom onset
  To further understand the underlying brain activity during post-stroke delirium we'll perform an additional electroencephalogram (EEG) to look at potential deviations in the brain activity that could be connected to this clinical presentation. We'll specifically look at the relative power in the beta frequency band.
The role of brain network disintegration in post-stroke delirium: electrical analysis of the relative power in the delta frequency band | first 72 hours after stroke symptom onset
  To further understand the underlying brain activity during post-stroke delirium we'll perform an additional electroencephalogram (EEG) to look at potential deviations in the brain activity that could be connected to this clinical presentation. We'll specifically look at the relative power in the delta frequency band.
The role of brain network disintegration in post-stroke delirium: electrical analysis of the relative power in the theta frequency band | first 72 hours after stroke symptom onset
  To further understand the underlying brain activity during post-stroke delirium we'll perform an additional electroencephalogram (EEG) to look at potential deviations in the brain activity that could be connected to this clinical presentation. We'll specifically look at the relative power in the theta frequency band.
The role of brain network disintegration in post-stroke delirium: electrical analysis of the relative power in the peak frequency band | first 72 hours after stroke symptom onset
  To further understand the underlying brain activity during post-stroke delirium we'll perform an additional electroencephalogram (EEG) to look at potential deviations in the brain activity that could be connected to this clinical presentation. We'll specifically look at the relative power in the peak frequency band.
The role of brain network disintegration in post-stroke delirium: electrical analysis of the phase lag index (PLI) | first 72 hours after stroke symptom onset
  To further understand the underlying brain activity during post-stroke delirium we'll perform an additional electroencephalogram (EEG) to look at potential deviations in the brain activity that could be connected to this clinical presentation. We'll specifically look at the phase lag index (PLI) to assess functional connectivity between time series based on the consistency with which one signal is leading or lagging with respect to another signal. The PLI characterizes the assymetry in the distribution of instantaneous phase differences between signals.
Post-stroke cognitive impairment | 3 months and 12 months after stroke symptom onset
  Using the Montreal Cognitive Assessment (MOCA) score. This is a maximum score of 30 points where a normal cognition is linked to a score of 26 or higher.
Post-stroke depression | 3 months and 12 months after stroke symptom onset
  Using the Patient Health Questionnaire-2 (PHQ-2). These scores range from 0 to 6. A score of 3 or higher indicates that major depressive disorder is likely.
Post-stroke depression | 3 months and 12 months after stroke symptom onset
  Using the Hospital Anxiety and Depression Scale (HADS). This test has a maximum of 21 points. Between 8 and 10 there is a possibility that the patient suffers from anxiety or depression. Between 11 and 21 it is likely that the patient suffers from anxiety or depression.
Markers of brain frailty | First 72 hours and 12 months after stroke symptom onset
  * visual rating of white matter hyperintensities using the Fazekas scale.
  * Visual rating of cerebral atrophy using the global cortical atrophy scale.

SECONDARY OUTCOMES:
Key drivers of post-stroke delirium. | 12 months after stroke symptom onset
  To determine if there are neuro-electrical key drivers of post-stroke delirium. We'll combine looking at impairment of functional brain connectivity strength and network disintegration.
Role infarct location | 12 months after stroke symptom onset
  To investigate the role of infarct location on development of post-stroke delirium. We'll analyse the anatomical location of the infarction to look if there is a connection betweet certain locations and the presence of post-stroke delirium in the patient.
Key drivers of post-stroke cognitive impairment. | 12 months after stroke symptom onset
  After determining if there is cognitive impairment, using the Montreal Cognitive Assessment (MOCA) score, we'll look at the electrical brain activity (both looking at persistent impairment of functional brain connectivity strength and network disintegration).

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No